CLINICAL TRIAL: NCT01960218
Title: Gas Exchange for Predicting Hospital Heart Failure Readmissions Clinical Evaluation Study
Brief Title: Gas Exchange for Predicting Hospital Heart Failure Readmissions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shape Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0512
Record Dates: First submitted 2013-10-04; First posted 2013-10-10 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: acute decompensated heart failure; gas exchange; cardiopulmonary; dyspnea; cardiopulmonary analyzer; heart disease; cardiovascular disease; cardiopulmonary exercise
MeSH Terms: conditions — Dyspnea; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute decompensated heart failure: Adult subjects anticipating discharge from a hospitalization where the primary discharge diagnosis is acute decompensated heart failure and who are not excluded due to existing conditions.

SUMMARY:
To determine whether, and if so, which gas exchange parameters measured on the Shape-HF Cardiopulmonary Exercise Testing System predict 30 and 180 day re-hospitalization in subjects discharged from hospitalization for an episode of acute decompensated heart failure.

DETAILED DESCRIPTION:
This is a prospective, single-specialty clinical study. This study is intended to evaluate the select gas exchange parameters during a short, sub-max bout of exercise using a simple stationary step on day of discharge to predict the subjects' readmission for acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 Years and older
* Subject is hospitalized for acute decompensated heart failure (ADHF)

  1. Systolic OR
  2. Diastolic
* Subject is Stage C:Class II/III/IV heart failure
* Subject is willing and to provide appropriate informed consent
* Subject is willing and able to comply with the requirements of the protocol, including follow-up evaluations and schedule
* Subject is willing to use the Shape-HF Cardiopulmonary Exercise Testing System

Exclusion Criteria:

* The subject is pregnant (verified in a manner consistent with institution's standard of care)
* Subject is currently participating in another investigational device or drug trial
* Subject is a prisoner, a minor or unable to adequately give informed consent due to mental or physical condition
* Subject is unwilling or unable to return for the required follow-up after test
* Subject has Left Ventricular Assist Device (LVAD)
* Subject is listed for transplant
* Subject has a clinical diagnosis of acute myocardial infarction (AMI) on admission (Note: If troponin measurements have been collected and are elevated but not due to an MI subject is still eligible for study)
* Subject has a pulmonary embolism (PE) on admission
* Subject is dialysis dependent
* Subject has a cardiac resynchronization device (CRT) which has been re-programmed at any time during the study
* Subject has Chronic Obstructive Pulmonary Disease (COPD) who is oxygen or steroid dependent
* Subject has severe hypertension > 180 millimeter of mercury (mmHg) resting systolic at time of test
* Subject has severe heart failure with renal insufficiency (with Creatinine clearance rate (CrCL) of 30 or less) and/or on IV Inotropic therapy and/or enrolling in hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be consecutively recruited from the population of subjects admitted to the hospital with acute decompensated heart failure.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-07 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
1. To evaluate if exercise gas exchange tests can predict 30 day hospital readmission for heart failure. | 30 days ± 3 days post discharge
  The analysis of exercise gas exchange (using the Shape-HF Cardiopulmonary Exercise Testing System) of the incidence of hospital readmission through 30 days ± 3 days post discharge follow-up.
2. To evaluate which gas exchange patterns were most highly associated with 30 day risk of readmission for recurrent acute decompensated heart failure. | 30 days ± 3 days post discharge
  The analysis of exercise gas exchange (using the Shape-HF Cardiopulmonary Exercise Testing System) of the incidence of hospital readmission through 30 days ± 3 days post discharge follow-up.
3. To determine the incidence of Adverse Events (AE) and Serious Adverse Events (SAE). | 30 days ± 3 days post discharge follow-up and through 180 days ± 15 days post discharge
  The analysis of the incidence of AEs and SAEs on the day of discharge post Shape-HF Cardiopulmonary Exercise Testing System through 30 days ± 3 days post discharge follow-up and through 180 days ± 15 days post discharge follow-up.

SECONDARY OUTCOMES:
1. To evaluate if exercise gas exchange tests can predict 180 day hospital readmission for heart failure. | 180 days ± 15 days post discharge
  The analysis of exercise gas exchange (using the Shape-HF Cardiopulmonary Exercise Testing System) of the incidence of hospital readmission through 180 days ± 15 days post discharge follow-up.
2. To evaluate which gas exchange patterns were most highly associated with 180 day risk of readmission for recurrent acute decompensated heart failure. | 180 days ± 15 days post discharge
  The analysis of exercise gas exchange (using the Shape-HF Cardiopulmonary Exercise Testing System) of the incidence of hospital readmission through 180 days ± 15 days post discharge follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham G Kocheril, MD, Principal Investigator — Christie Clinc
Locations (7):
- United States (7):
  - Veterans Affairs-Washington DC, Washington D.C., District of Columbia
  - Christie Clinic, Champaign, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fairview Southdale, Edina, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Background] Fang J, Mensah GA, Croft JB, Keenan NL. Heart failure-related hospitalization in the U.S., 1979 to 2004. J Am Coll Cardiol. 2008 Aug 5;52(6):428-34. doi: 10.1016/j.jacc.2008.03.061. PMID 18672162
- [Background] Pulignano G, Del Sindaco D, Tavazzi L, Lucci D, Gorini M, Leggio F, Porcu M, Scherillo M, Opasich C, Di Lenarda A, Senni M, Maggioni AP; IN-CHF Investigators. Clinical features and outcomes of elderly outpatients with heart failure followed up in hospital cardiology units: data from a large nationwide cardiology database (IN-CHF Registry). Am Heart J. 2002 Jan;143(1):45-55. doi: 10.1067/mhj.2002.119608. PMID 11773911
- [Background] Jacobs B. Reducing heart failure hospital readmissions from skilled nursing facilities. Prof Case Manag. 2011 Jan-Feb;16(1):18-24; quiz 25-6. doi: 10.1097/NCM.0b013e3181f3f684. PMID 21164330
- [Background] Yu CM, Wang L, Chau E, Chan RH, Kong SL, Tang MO, Christensen J, Stadler RW, Lau CP. Intrathoracic impedance monitoring in patients with heart failure: correlation with fluid status and feasibility of early warning preceding hospitalization. Circulation. 2005 Aug 9;112(6):841-8. doi: 10.1161/CIRCULATIONAHA.104.492207. Epub 2005 Aug 1. PMID 16061743